CLINICAL TRIAL: NCT03944109
Title: The Safety, Tolerability and Efficacy of Multiple Subcutaneous Injections of SHR-1209 in Subjects With Hyperlipidemia - A PhaseⅠb/Ⅱ Randomized, Double-Blind, Placebo-Controlled Clinical Study
Brief Title: The Safety, Tolerability and Efficacy of Multiple Subcutaneous Injections of SHR-1209 in Subjects With Hyperlipidemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR-1209-102
Record Dates: First submitted 2019-05-04; First posted 2019-05-09 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-07

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1209 (Experimental): Participants received one of 6 dose levels of SHR-1209 administered as multiple subcutaneous doses.
  Interventions: Drug: SHR-1209
- Placebo (Placebo Comparator): Participants received matching placebo dose regimens by subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1209 — Pharmaceutical form: lyophilized formulation
  Route of administration: subcutaneous
  Arms: SHR-1209
Drug: Placebo — Pharmaceutical form: lyophilized formulation
  Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo- controlled phaseⅠb/Ⅱclinical study. Totally 108 subjects are planned to enrolled with 36 subjects in three low-dose groups (group 1, group 2 and group 3) and 72 subjects in three high-dose groups (group 4, group 5, and group 6).12 subjects with hyperlipidemia who received statin stable treatment for more than 28 days are enrolled in each low-dose group, randomly given SHR-1209 or placebo treatment at a ratio of 5:1. 24 subjects with hyperlipidemia who received statin stable treatment for more than 28 days are enrolled in each high-dose group, randomly given SHR-1209 or placebo treatment at a ratio of 5:1. The primary objective of this study is to evaluate the safety, tolerability, and efficacy of multiple subcutaneous injections of SHR-1209 in hyperlipidemia subjects treated with stabilized dose of statin. Groups detail as follows:

1. SHR-1209 dose 1 /placebo frequence 1
2. SHR-1209 dose 2 /placebo frequence 2
3. SHR-1209 dose 3 /placebo frequence 3
4. SHR-1209 dose 4 /placebo frequence 1
5. SHR-1209 dose 5 /placebo frequence 2
6. SHR-1209 dose 6 /placebo frequence 3

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤65 years old;
2. Subjects who are receiving statin therapy at the time of screening or who are eligible for statin therapy can randomized to receive a stable dose of statin therapy for more than 28 days and are willing to maintain stable statin therapy in this study;
3. Low-density lipoprotein cholesterol (LDL-C) level ≥2.6mmol/L of subjects who receiving statin and/or other lipid-lowering therapy at the time of screening, or LDL-C≥ 3.4mmol/L of subjects who didn't receive any-lowering therapy at the time of screening, and LDL-C still ≥2.6mmol/L before randomization;
4. Fasting triglycerides ≤4.5 mmol/L;
5. Body mass index (BMI) ≥18 and ≤ 35 kg/m2;
6. Signed informed consent.

Exclusion Criteria:

1. A clinical history of drug allergy or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known allergy to experimental or similar experimental drugs;
2. Diagnosis of homozygous familial hypercholesterolemia;
3. New York heart association (NYHA) defined Ⅱ - Ⅳ history of heart failure;
4. History of acute coronary syndrome (e.g. myocardial infarction, hospitalization for unstable angina), or percutaneous coronary intervention, or coronary artery bypass graft, or history of cerebrovascular disease, within 12 months prior to screening;
5. Uncontrolled severe arrhythmias that are not controlled by drugs or other therapy within 12 months prior to enrollment;
6. Uncontrolled hypertension (systolic blood pressure ≥ 160 and/or diastolic blood pressure ≥ 100 mmHg);
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma pancreatic acyl transferase (GGT), more than 2.5x ULN;
8. Subjects with previous malignant tumor diseases. etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Primary efficacy end point:Percent change from baseline to end of the dosing interval in LDL-C. | Baseline to day 113 for group1,2,4,5 or day 169 for group 3,6
Primary safety end point:Number of subjects with adverse events. | Baseline to day 169 for group 1,3,4,6 or day 141 for group 2,5

SECONDARY OUTCOMES:
Absolute change from baseline to end of the dosing interval in LDL-C. | Baseline to day 113 for group1,2,4,5 or day 169 for group 3,6
Percent change from baseline to day 85 in LDL-C. | Baseline to day 85 for all 6 groups
Absolute change from baseline to day 85 in LDL-C. | Baseline to day 85 for all 6 groups
Percent change in PCSK9. | Baseline to day 169 for group 1,3,4,6 or day 141 for group 2,5
Absolute change in PCSK9. | Baseline to day 169 for group 1,3,4,6 or day 141 for group 2,5

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital ,The Second Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053
- [Derived] Xu M, Zhu X, Wu J, Zhang Y, Zhao D, Wang X, Ding Y, Cao Y, Li C, Hu W, Sheng J, Luo Z, Zheng Z, Hu J, Liu J, Zhou X, Shen A, Ding X, Zhang Y, Zhao Y, Li Y, Zhong S, An S, Zou J, Yan L. PCSK9 inhibitor recaticimab for hypercholesterolemia on stable statin dose: a randomized, double-blind, placebo-controlled phase 1b/2 study. BMC Med. 2022 Jan 18;20(1):13. doi: 10.1186/s12916-021-02208-w. PMID 35039035